CLINICAL TRIAL: NCT02864394
Title: A Multinational, Multicenter, Phase III, Randomized Open-label Trial of Pembrolizumab Versus Docetaxel in Previously Treated Subjects With Non-Small Cell Lung Cancer
Brief Title: Study of Pembrolizumab Versus Docetaxel in Participants Previously Treated for Non-Small Cell Lung Cancer (MK-3475-033/KEYNOTE-033)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-033; MK-3475-033 (Other: Merck Registration Number); KEYNOTE-033 (Other: MSD)
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants with NSCLC receive pembrolizumab 2 mg/kg intravenously (IV) over 30 minutes every 3 weeks (Q3W) for up to 35 doses (approximately 24 months).
  Interventions: Biological: Pembrolizumab
- Docetaxel (Experimental): Participants with NSCLC receive Docetaxel 75 mg/m^2 IV over 1 hour Q3W until disease progression, toxicity, investigator's decision to discontinue, or consent withdrawal.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab administered IV at 2 mg/kg on Day 1 of each 21-day cycle for up to 35 doses (approximately 24 months).
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: Docetaxel — Docetaxel administered IV at 75 mg/m^2 on Day 1 of each 21-day cycle as per the approved product label.
  Other Names: TAXOTERE®
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to assess the efficacy of pembrolizumab (MK-3475) versus docetaxel in participants with non-small cell lung cancer (NSCLC) with programmed cell death ligand 1 (PD-L1) positive tumors who have experienced disease progression after platinum-containing systemic therapy. The primary hypotheses of this study are that pembrolizumab (MK-3475) prolongs overall survival (OS) and that pembrolizumab prolongs progression-free survival (PFS), compared to docetaxel in participants with PD-L1 positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants must be born, raised, and reside in China
* Has a histologically or cytologically confirmed diagnosis of stage IIIB/IV or recurrent NSCLC and have at least one measurable lesion as defined by RECIST 1.1
* Has a life expectancy of ≥3 months
* Has progression of disease (investigator determined) per RECIST 1.1 after treatment with at least two cycles of a platinum-containing doublet
* Has documentation of epidermal growth factor receptor (EGFR) mutation and anaplastic lymphoma kinase (ALK) translocation status
* Participants with an EGFR sensitizing mutation tumor will be excluded
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 within 10 days prior to study start
* Has provided archival tumor tissue sample or newly obtained formalin fixed tumor tissue from a recent biopsy of a tumor lesion not previously irradiated
* Has a PD-L1 positive tumor as determined by immunohistochemistry at a central laboratory
* Has resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia)
* Has recovered from the toxicity and/or complications of any recent major surgery or radiation therapy
* Females must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours prior to receiving the first dose of study medication)
* Female and male participants of reproductive potential must agree to use adequate contraception starting with the first dose of study therapy through 120 days after the last dose of pembrolizumab (MK-3475) or 180 days after the last dose of docetaxel

Exclusion Criteria:

* Has received prior therapy with docetaxel for NSCLC
* Is currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment
* Is receiving systemic steroid therapy within 3 days prior to the first dose of study treatment or receiving any other form of immunosuppressive
* Is expected to require any other form of systemic or localized antineoplastic therapy while on study including maintenance therapy with another agent for NSCLC or radiation therapy
* Has received prior systemic cytotoxic chemotherapy, antineoplastic biological therapy (e.g., cetuximab), any other agents used as systemic treatment for cancer, or major surgery within 3 weeks of the first dose of study treatment; received thoracic radiation therapy of > 30 Gray Units (Gy) within 6 months of the first dose of study treatment; received prior ALK-directed tyrosine kinase inhibitor therapy or completed palliative radiotherapy of 30 Gy or less within 7 days of the first dose of study treatment
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-PD-L1, anti-PD-L2, with an agent directed to an agonist or antagonist T-cell check point receptor, or if the participant has previously participated in Merck sponsored clinical trials evaluating pembrolizumab (MK-3475)
* Has a known additional malignancy that is progressing or requires active treatment, with the exception of early stage cancers, treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in past 2 years
* Has had an allogeneic tissue/solid organ transplant
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has received or will receive a live vaccine within 30 days prior to the first administration of study medication
* Has an active infection requiring intravenous systemic therapy
* Has known history of Human Immunodeficiency Virus (HIV) (HIV ½ antibodies)
* Has known active Hepatitis B or C
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Is pregnant or breastfeeding, or expecting to conceive or father children starting with the screening visit (Visit 1) through 120 days after the last dose of pembrolizumab (MK-3475) or 180 days after the last dose of docetaxel
* Requires treatment with a strong inhibitor of Cytochrome P450 3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ren S, Feng J, Ma S, Chen H, Ma Z, Huang C, Zhang L, He J, Wang C, Zhou J, Danchaivijtr P, Wang CC, Vynnychenko I, Wang K, Orlandi F, Sriuranpong V, Li B, Ge J, Dang T, Zhou C. KEYNOTE-033: Randomized phase 3 study of pembrolizumab vs docetaxel in previously treated, PD-L1-positive, advanced NSCLC. Int J Cancer. 2023 Aug 1;153(3):623-634. doi: 10.1002/ijc.34532. Epub 2023 May 4. PMID 37141294
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26058&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with non-small cell lung cancer (NSCLC) and programmed cell death ligand 1 (PD-L1) positive (Tumor Proportion Score [TPS] ≥1%) tumors who had experienced disease progression after platinum-containing systemic therapy were recruited.
Pre-assignment Details: Of 425 participants randomized, 411 received treatment on study. All 425 participants were PD-L1 positive (TPS ≥1%). At the time of the Final Analysis data cut-off (09-Sep-2019), 130 participants were ongoing in the study. No participants were ongoing in the study as of the final adverse event collection date (14-Oct-2022).
Period: Overall Study
Arm/Group | Pembrolizumab | Docetaxel
Started | 213 | 212
Treated | 213 | 198
Received Second Course Pembrolizumab Treatment | 10 | 0
Completed | 0 | 0
Not Completed | 213 | 212
Not completed — Death | 184 | 189
Not completed — Lost to Follow-up | 0 | 2
Not completed — Sponsor Decision | 26 | 11
Not completed — Withdrawal by Subject | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Docetaxel | Total
Number analyzed (Participants) | 213 | 212 | 425
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (8.8) | 61.0 (9.2) | 60.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 48 | 104
  Male | 157 | 164 | 321
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 198 | 198 | 396
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 181 | 177 | 358
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 32 | 35 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
PD-L1 Status [Count of Participants; unit: Participants] — Participants were stratified by extent of tumoral PD-L1 expression (TPS 1-49% vs. TPS ≥50%).
  Participants
    TPS ≥50% | 114 | 112 | 226
    TPS = 1-49% | 98 | 98 | 196
    TPS <1% | 0 | 2 | 2
    NOT EVALUABLE | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Positive (Tumor Proportion Score [TPS] ≥50%) Tumors
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS was reported by treatment arm for participants in the TPS ≥50% stratum of PD-L1 expression.
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥50%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 114 | 113
Months | 12.3 [10.0 to 16.3] | 10.9 [8.3 to 13.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; Treatment comparison (Hazard Ratio, HR) based on Cox regression model with Efron's method of tie handling with treatment as a covariate. One-sided p-value was based on log-rank test; Test type: Superiority; p = 0.1276, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.61 to 1.14]

2. Primary Outcome: OS in Participants With PD-L1 Positive (TPS ≥1%) Tumors (All Participants)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS was reported by treatment arm for participants in the TPS ≥1% stratum of PD-L1 expression (all participants).
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥1% (all participants).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 212
Months | 12.9 [10.3 to 16.5] | 10.6 [8.7 to 12.5]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; OS was not formally tested. Treatment comparison (HR) based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by PD-L1 expression status (TPS ≥50% vs. TPS 1-49%). A nominal one-sided p-value for testing was based on log-rank test stratified by PD-L1 expression status (TPS ≥50% vs. TPS 1-49%); Test type: Other; p = 0.0076, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.95]

3. Primary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With PD-L1 Positive (TPS ≥50%) Tumors
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, PFS was reported by treatment arm for participants in the TPS ≥50% stratum of PD-L1 expression.
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥50%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 114 | 113
Months | 4.0 [2.1 to 8.0] | 2.5 [2.1 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; PFS was not formally tested. Treatment comparison (HR) based on Cox regression model with Efron's method of tie handling with treatment as a covariate. A nominal one-sided p-value for testing was based on log-rank test; Test type: Other; p = 0.0534, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.54 to 1.07]

4. Primary Outcome: PFS Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 Positive (TPS ≥1%) Tumors (All Participants)
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the SOD of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, PFS was reported by treatment arm for participants in the TPS ≥1% stratum of PD-L1 expression (all participants).
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥1% (all participants).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 212
Months | 3.3 [2.1 to 4.1] | 3.0 [2.3 to 4.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; PFS was not formally tested. Treatment comparison (HR) based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by PD-L1 expression status (TPS ≥50% vs. TPS 1-49%). A nominal one-sided p-value for testing was based on log-rank test stratified by PD-L1 expression status (TPS ≥50% vs. TPS 1-49%); Test type: Other; p = 0.0847, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.08]

5. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 Positive (TPS ≥50%) Tumors
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by BICR. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for participants in the TPS ≥50% stratum of PD-L1 expression.
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥50%
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 114 | 113
Percentage of Participants | 28.1 [20.1 to 37.3] | 7.1 [3.1 to 13.5]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; ORR was not formally tested. Treatment comparison was based on the Miettinen & Nurminen method. A nominal one-sided p-value for testing was calculated; Test type: Other; p < 0.0001, Miettinen & Nurminen Method; Difference in Percentage = 21.0, 95% CI 2-sided [11.5 to 30.7]

6. Secondary Outcome: ORR Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 Positive (TPS ≥1%) Tumors (All Participants)
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by BICR. Per protocol, the percentage of participants who experienced CR or PR is reported here as the ORR for participants in the TPS ≥1% stratum of PD-L1 expression (all participants).
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants with PD-L1 TPS ≥1% (all participants).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 212
Percentage of Participants | 20.7 [15.4 to 26.7] | 5.7 [3.0 to 9.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Docetaxel; ORR was not formally tested. Treatment comparison was based on Miettinen & Nurminen method stratified by PD-L1 expression status (TPS>=50% vs. TPS 1-49%). If no participants were in one of the treatment arms involved in a comparison for a particular stratum, then that stratum was excluded from the treatment comparison. A nominal one-sided p-value for testing was calculated; Test type: Other; p < 0.0001, Miettinen & Nurminen Method; Difference in Percentage = 15.0, 95% CI 2-sided [8.8 to 21.6]

7. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 Positive (TPS ≥50%) Tumors
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The appearance of one or more new lesions was also considered PD. Response duration was calculated using the Kaplan-Meier method for censored data. Per protocol, DOR was reported by treatment arm for participants in the TPS ≥50% stratum of PD-L1 expression.
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants in the PD-L1 TPS ≥50% stratum who demonstrated a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 32 | 8
Months | 16.6 [10.0 to NA] — NA = Upper limit of 95% confidence interval not reached at time of data cut-off due to insufficient number of responding participants with relapse | 6.4 [4.1 to NA] — NA = Upper limit of 95% confidence interval not reached at time of data cut-off due to insufficient number of responding participants with relapse

8. Secondary Outcome: DOR Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 Positive (TPS ≥1%) Tumors (All Participants)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Response duration was calculated using the Kaplan-Meier method for censored data. Per protocol, DOR was reported by treatment arm for participants in the TPS ≥1% stratum of PD-L1 expression (all participants).
Time Frame: Up to approximately 36 months (through Final Analysis cut-off date of 09-Sep-2019)
Population: All randomized participants in the PD-L1 TPS ≥1% stratum who demonstrated a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 44 | 12
Months | 16.6 [10.2 to NA] — NA = Upper limit of 95% confidence interval not reached at time of data cut-off due to insufficient number of responding participants with relapse | 6.3 [3.9 to NA] — NA = Upper limit of 95% confidence interval not reached at time of data cut-off due to insufficient number of responding participants with relapse

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the study intervention are excluded. Per protocol, the number of participants who experienced an AE was reported by treatment arm for all participants as part of the pre-specified safety analysis at study completion (Final AE collection cut-off date of 14-Oct-2022).
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 198
Participants | 206 | 187

10. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Per protocol, the number of participants who discontinued study treatment due to an AE was reported by treatment arm for all participants as part of the pre-specified safety analysis at study completion (Final AE collection cut-off date of 14-Oct-2022).
Time Frame: Up to approximately 45 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 198
Participants | 32 | 24

11. Secondary Outcome: Number of Participants Who Experienced an Adverse Event of Special Interest (AEOSI)
Description: An AEOSI was defined as any AE that is immune-mediated or potentially immune-mediated. An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Per protocol, the number of participants who experienced an AE was reported by treatment arm for all participants as part of the pre-specified safety analysis at study completion (Final AE collection cut-off date of 14-Oct-2022).
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 198
Participants | 63 | 12

12. Secondary Outcome: Number of Participants Who Experienced a Grade 3-5 AE
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the study intervention are excluded. Per protocol, the number of participants who experienced an AE was reported by treatment arm for all participants as part of the pre-specified safety analysis at study completion (Final AE collection cut-off date of 14-Oct-2022).
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 198
Participants | 86 | 117

13. Secondary Outcome: Number of Participants Who Experienced an AE That Was Experienced by ≥10% of Participants in Either Arm
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition temporally associated with the use of the Sponsor's product was also an AE. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the study intervention are excluded. Per protocol, the number of participants who experienced an AE was reported by treatment arm for all participants (TPS ≥1% stratum of PD-L1 expression) as part of the pre-specified safety analysis at study completion (Final AE collection cut-off date of 14-Oct-2022).
Time Frame: Up to approximately 66 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Docetaxel
Number analyzed (Participants) | 213 | 198
Participants | 206 | 187

ADVERSE EVENTS:
Time Frame: Up to approximately 66 months
Description: All-Cause Mortality table includes all randomized participants.
  Serious and Other AEs include all randomized participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug were excluded as AEs.
Groups:
- Pembrolizumab: Participants with NSCLC receive pembrolizumab 2 mg/kg intravenously (IV) over 30 minutes Q3W for up to 35 doses (approximately 24 months).
- Pembrolizumab 2ⁿᵈ Course: Following treatment response, participants from the "Pebrolizumab" arm could opt to receive pembrolizumab 2 mg/kg intravenously (IV) over 30 minutes Q3W for up to 17 additional doses, if they met protocol-specific criteria.
Arm/Group | Pembrolizumab | Docetaxel | Pembrolizumab 2ⁿᵈ Course
All-Cause Mortality (participants affected / at risk) | 182/213 | 195/212 | 3/10
Serious Adverse Events (participants affected / at risk) | 77/213 | 75/198 | 2/10
Other Adverse Events (participants affected / at risk) | 193/213 | 182/198 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=213) | Docetaxel (N=198) | Pembrolizumab 2ⁿᵈ Course (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 17 (18) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 13 (21) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Paratyphoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 24 (25) | 19 (21) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglossal nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=213) | Docetaxel (N=198) | Pembrolizumab 2ⁿᵈ Course (N=10)
Anaemia (Blood and lymphatic system disorders) | 71 (100) | 93 (151) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 5 (10) | 35 (65) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (6) | 48 (83) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 21 (22) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 28 (37) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (24) | 25 (31) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 19 (26) | 32 (43) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (16) | 35 (83) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (21) | 20 (29) | 0 (0)
Asthenia (General disorders) | 20 (20) | 31 (37) | 1 (1)
Chest discomfort (General disorders) | 6 (6) | 7 (7) | 1 (1)
Chest pain (General disorders) | 27 (34) | 16 (17) | 0 (0)
Fatigue (General disorders) | 22 (26) | 37 (42) | 0 (0)
Malaise (General disorders) | 14 (16) | 8 (11) | 0 (0)
Oedema peripheral (General disorders) | 7 (7) | 19 (25) | 0 (0)
Pyrexia (General disorders) | 22 (32) | 21 (24) | 2 (3)
Pneumonia (Infections and infestations) | 25 (26) | 14 (14) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 18 (26) | 5 (6) | 0 (0)
Alanine aminotransferase increased (Investigations) | 38 (54) | 15 (19) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 46 (61) | 14 (16) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 21 (22) | 4 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 16 (31) | 5 (9) | 1 (1)
Blood cholesterol increased (Investigations) | 19 (33) | 13 (14) | 0 (0)
Blood creatinine increased (Investigations) | 13 (25) | 5 (8) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 6 (6) | 1 (1) | 2 (2)
Blood triglycerides increased (Investigations) | 13 (43) | 9 (19) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 21 (29) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (7) | 28 (84) | 0 (0)
Platelet count decreased (Investigations) | 9 (19) | 6 (7) | 1 (1)
Prealbumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 45 (52) | 25 (26) | 1 (1)
Weight increased (Investigations) | 11 (19) | 3 (3) | 0 (0)
White blood cell count decreased (Investigations) | 5 (5) | 54 (132) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 42 (54) | 51 (62) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 22 (46) | 9 (13) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 18 (30) | 8 (9) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 11 (24) | 6 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 45 (57) | 38 (45) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (16) | 5 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 26 (33) | 19 (24) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 25 (33) | 15 (19) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 13 (24) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (27) | 17 (26) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (25) | 18 (19) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 11 (18) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (16) | 16 (21) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 13 (14) | 0 (0)
Insomnia (Psychiatric disorders) | 28 (32) | 24 (31) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (56) | 29 (31) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 (42) | 32 (38) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 34 (53) | 19 (24) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 10 (11) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 93 (97) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (27) | 5 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 35 (55) | 14 (18) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Protocol amendment 5 called for participant discontinuation from this study under protocol-specified circumstances.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT02864394/Prot_SAP_001.pdf